CLINICAL TRIAL: NCT04311996
Title: Does Social Buffering Continue to be Effective Over the Peripubertal Period When Friends Share the Stressor Experience?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00006378-3
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Adolescent Behavior; Social Stress
MeSH Terms: conditions — Adolescent Behavior | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Friend and Target Both (Experimental): There are four conditions: (1) Friend and Target both undergo the stressor, (2) Friend provides support but does not undergo the stressor, (3) Unfamiliar Peer and Target undergo the stressor, and (4) Alone (no partner).
  Interventions: Other: Friend and target
- Experimental: Friend Provides Support (Experimental): There are four conditions: (1) Friend and Target both undergo the stressor, (2) Friend provides support but does not undergo the stressor, (3) Unfamiliar Peer and Target undergo the stressor, and (4) Alone (no partner).
  Interventions: Other: Friend support
- Experimental: Unfamiliar Peer and Target (Experimental): There are four conditions: (1) Friend and Target both undergo the stressor, (2) Friend provides support but does not undergo the stressor, (3) Unfamiliar Peer and Target undergo the stressor, and (4) Alone (no partner).
  Interventions: Other: unfamiliar peer and target
- Experimental: Alone (Experimental): There are four conditions: (1) Friend and Target both undergo the stressor, (2) Friend provides support but does not undergo the stressor, (3) Unfamiliar Peer and Target undergo the stressor, and (4) Alone (no partner).
  Interventions: Other: alone

INTERVENTIONS:
Other: Friend and target — random assignment to Friend and Target Both condition
  Arms: Experimental: Friend and Target Both
Other: Friend support — random assignment to Friend Provides Support condition
  Arms: Experimental: Friend Provides Support
Other: unfamiliar peer and target — random assignment to Unfamiliar Peer and Target condition
  Arms: Experimental: Unfamiliar Peer and Target
Other: alone — random assignment to Alone condition
  Arms: Experimental: Alone

SUMMARY:
The purpose of this experiment is to determine whether social buffering by friends of stress physiology remains effective later in puberty when friends share the load versus when they provide support but are not undergoing the stressor with the target child. There are four conditions: (1) Friend and Target both undergo the stressor, (2) Friend provides support but does not undergo the stressor, (3) Unfamiliar Peer and Target undergo the stressor, and (4) Alone (no partner).

DETAILED DESCRIPTION:
Adolescents experience social evaluation stress frequently. However, it is likely that often they are not alone, but with friends who are also going through the same experience. Thus, it is possible that under these conditions, social buffering by friends does not wane over the peripubertal period. Participants will be assigned to social conditions while engaging in an evaluative stressor task.

ELIGIBILITY:
Inclusion Criteria:

* sufficient vision, hearing, and language skills to provide verbal and written assent
* ability to see and read stimuli presented on the computer screen
* ability to hear verbal instructions provided by the experimenter and judges

Exclusion Criteria:

* premature birth (less than 37 weeks)
* congenital and/or chromosomal disorders (e.g. cerebral palsy, FAS, mental retardation, Turner Syndrome, Down Syndrome, Fragile X)
* Autism Spectrum Disorders
* history of serious medical illness (e.g., cancer, organ transplant)
* serious psychiatric illness
* systemic glucocorticoids or beta-adrenergic medication use

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 269 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan Gunnar, PhD, Principal Investigator — University of Minnesota; Kathleen Thomas, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Friend and Target Both: Friend Also social buffer: Target experiences TSST stressor with a friend who also experiences the stressor
- Experimental: Friend Provides Support: Friend Support social buffer: Target experiences TSST stressor with a friend who does NOT experience the stressor
- Experimental: Unfamiliar Peer and Target: Unfamiliar Peer social buffer: Target experiences TSST stressor with an unfamiliar peer who also experiences the stressor
- Experimental: Alone: no social buffer: random assignment to Alone Condition, where Target experiences the TSST alone
Period: Overall Study
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Started | 63 | 72 | 65 | 69
Completed | 61 | 65 | 62 | 68
Not Completed | 2 | 7 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone | Total
Number analyzed (Participants) | 61 | 65 | 62 | 68 | 256
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 65 | 62 | 68 | 256
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.98 (1.05) | 12.98 (1.05) | 12.94 (0.91) | 13.15 (1.11) | 13.02 (1.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 33 | 31 | 32 | 127
  Male | 30 | 32 | 31 | 36 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 5 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 47 | 54 | 55 | 57 | 213
  More than one race | 10 | 7 | 1 | 6 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cortisol AUCi
Description: Cortisol response to the TSST, measured as Area Under the Curve, increase from baseline. 7 Samples were taken during the course of the assessment, at (1) arrival for training purposes; (2) after the calming video, 30 minutes after arrival; (3) after 5 minutes of speech preparation; (4) after 10+minutes of speech and math performance; (5) 15 minutes after sample 4; (6) 10 minutes after sample 5; (7) 10 minutes after sample 6. Area under the curve at intercept (AUCi) is calculated using samples 2-7 with sample 2 as the intercept.
Time Frame: 2 hours
Population: 256 participants were completed, with 61 Friend and Target Both, 65 Friend Support, 62 Unfamiliar Peer, and 68 Alone. For each outcomes, all available analyzable data were included in results, sometimes resulting in lower n.
Measure: Mean (Standard Deviation); unit: (ug/dl)*minutes
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 63 | 61 | 66
(ug/dl)*minutes | 0.0043 (0.06) | 0.0256 (0.06) | 0.0177 (0.05) | 0.022 (0.06)

2. Primary Outcome: sAA AUCi
Description: Salivary Alpha Amylase response to the TSST, measured as Area Under the Curve, increase from baseline. 7 Samples were taken during the course of the assessment, at (1) arrival for training purposes; (2) after the calming video, 30 minutes after arrival; (3) after 5 minutes of speech preparation; (4) after 10+minutes of speech and math performance; (5) 15 minutes after sample 4; (6) 10 minutes after sample 5; (7) 10 minutes after sample 6. Of those, samples (2, 4, 5) are assayed for salivary alpha amylase (sAA) in micrograms per milliliter. Area under the curve at intercept (AUCi) is calculated using samples 2, 4, 5 with sample 2 as the intercept.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: (ug/mL)*minute
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 53 | 56 | 55 | 65
(ug/mL)*minute | 0.0364 (0.12) | 0.0434 (0.09) | 0.0021 (0.14) | 0.0255 (0.08)

3. Secondary Outcome: Self Report of Stress
Description: Self-report of stress using a Likert-type scale with 5 levels of stress felt: (1) Not At All, (2) A Little, (3) Some, (4) A Lot, (5) A Whole Lot. Level of stress was reported for at these points during the assessment: (1) How stressed did you feel when you first connected on the video call and saw the experimenter?, (2) How stressful was the period of time before we started the video?, (3) How stressful did you feel while watching the video?, (4) How stressful was the period of time when you were preparing your speech and thinking about what to say?, (5) How stressful was giving the speech?, (6) How stressful was the math portion?, (7) How stressed do you feel now, after the speech and math portions are done? Self reported stress was computed as the mean of items (4, 5, 6) - item 1.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 67
score on a scale | 1.65 (0.86) | 1.6 (1.02) | 1.65 (0.99) | 1.79 (0.97)

4. Other Pre Specified Outcome: Hours Since Awakening. Potential Covariate
Description: Participants report the number of hours between waking up on the day of assessment and the start of the TSST test.
  This is only a potential covariate for cortisol, which follows a circadian rhythm.
Time Frame: day of testing session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 68
hours | 8.45 (2.03) | 7.8 (2.04) | 8.26 (2.06) | 8.59 (1.87)

5. Other Pre Specified Outcome: Pretax Family Income. Potential Covariate
Description: Parents report on gross family income on an 11-point ordinal scale: (1) Less than $15,000, (2) $15,001 to $25,000, (3) $25,001 to $35,000, (4) $35,001 to $50,000, (5) $50,001 to $75,000, (6) $75,001 to $100,000, (7) $100,001 to $125,000, (8) $125,001 to $150,000, (9) $150,001 to $175,000, (10) $175,001 to 200,000, (11) $200,001 or more
Time Frame: calendar year previous to TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 60 | 64 | 58 | 67
score on a scale | 9 (2.37) | 9 (1.98) | 8 (2.04) | 9 (2.18)

6. Other Pre Specified Outcome: Parental Average Education Level. Potential Covariate
Description: Parents report education level for both parents on a 6-point ordinal scale: (1) Less than high school degree, (2) High school or GED, (3) Associate degree, college academia program, (4) Bachelor's degree, (5) Master's degree, (6) Professional and/or Doctorate degree. Average of parents' education is calculated and reported.
Time Frame: lifetime
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 68
score on a scale | 4.5 (0.78) | 4.5 (0.87) | 4.5 (0.78) | 4.5 (0.72)

7. Other Pre Specified Outcome: Number of Adults in the Home. Potential Covariate
Description: Parents report on how many adults are living in the home.
Time Frame: day of TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: persons
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 68
persons | 1.97 (0.36) | 1.97 (0.47) | 1.95 (0.34) | 2 (0.42)

8. Other Pre Specified Outcome: Caffeine or Nicotine Use. Potential Covariate
Description: Youth report on whether they consumed caffeine or nicotine in the 1-2 hours prior to the TSST assessment. Coded as no=0, yes=1. Used as a potential covariate for heart rate and neuroendocrine measures.
Time Frame: 1-2 hours prior to TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 66
score on a scale | 0.05 (0.22) | 0.02 (0.13) | 0.06 (0.25) | 0.05 (0.21)

9. Other Pre Specified Outcome: Granger Score. Potential Covariate
Description: The Granger score (ordinal, modeled continuously) is a score based on work by Doug Granger of medications that can affect activity of the HPA axis, weighted by significance of potential impact (Granger, Hibel, Fortunato, & Kapelewski, 2009). Each medication taken is given a score of 0, 1, or 2, and all medication scores for a participant is summed, resulting in scores from 0 to infinity. Lower scores are less likely to influence cortisol. Potential Covariate
Time Frame: day of 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 67
score on a scale | 0.34 (0.83) | 0.28 (0.79) | 0.19 (0.6) | 0.64 (1.36)

10. Other Pre Specified Outcome: Quality of Relationship With Primary Parent, BSV Positive Attachment Scale. Potential Covariate
Description: Network of Relationships Inventory (NRI) reported by youth for their primary parent on how much they experience various emotions or incidents (e.g. How much free time do you spend with this person?), reported on a 5-point scale: (1) Little or None, (2) Somewhat, (3) Very Much, (4) Extremely Much, (5) The Most. Mean scores calculated from all positive attachment items, range 1-5. Potential Covariate. This self report reflects the general current state of the relationship, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 66
score on a scale | 3.22 (0.74) | 3.44 (0.79) | 3.23 (0.7) | 3.26 (0.85)

11. Other Pre Specified Outcome: Quality of Relationship With Close Friend, BSV Positive Attachment Scale. Potential Covariate
Description: Network of Relationships Inventory (NRI) reported by youth for their close friend on how much they experience various emotions or incidents (e.g. How much free time do you spend with this person?), reported on a 5-point scale: (1) Little or None, (2) Somewhat, (3) Very Much, (4) Extremely Much, (5) The Most. Mean scores calculated from all positive attachment items, ranging 1-5. Potential Covariate. This self report reflects the general current state of the relationship, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 64 | 62 | 66
score on a scale | 3.18 (0.71) | 3.36 (0.71) | 3.31 (0.73) | 3.27 (0.73)

12. Other Pre Specified Outcome: Peer Acceptance/Rejection. Potential Covariate
Description: Scale on the MacArthur Health and Behavior Questionnaire, 5pt scale (1-5), high scores indicate peer acceptance. This report reflects the general current state of the youth, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 68
score on a scale | 3.61 (0.69) | 3.62 (0.41) | 3.67 (0.31) | 3.56 (0.41)

13. Other Pre Specified Outcome: Behavioral Inhibition. Potential Covariate
Description: Scale on the MacArthur Health and Behavior Questionnaire, 3pt scale (0,1,2), high scores indicate inhibition. This report reflects the general current state of the youth, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 68
score on a scale | 0.69 (0.62) | 0.52 (0.43) | 0.64 (0.54) | 0.69 (0.51)

14. Other Pre Specified Outcome: Internalizing Symptoms. Potential Covariate
Description: Higher order measure from the MacArthur Health and Behavior Questionnaire, 3pt scale (0,1,2), high scores indicate Internalizing. This report reflects the general current state of the youth, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 66
score on a scale | 0.26 (0.17) | 0.24 (0.22) | 0.25 (0.2) | 0.26 (0.22)

15. Other Pre Specified Outcome: Externalizing Symptoms. Potential Covariate
Description: Higher order measure from the MacArthur Health and Behavior Questionnaire, 3pt scale (0,1,2), high scores indicate externalizing. This report reflects the general current state of the youth, without a specific timeframe, and was obtained during the TSST session.
Time Frame: 2 hour TSST session
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Friend and Target Both | Experimental: Friend Provides Support | Experimental: Unfamiliar Peer and Target | Experimental: Alone
Number analyzed (Participants) | 61 | 65 | 62 | 67
score on a scale | 0.11 (0.13) | 0.13 (0.13) | 0.14 (0.15) | 0.14 (0.16)

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Friend and Target Both: random assignment to Friend and Target Condition, where both undergo stressor
  Friend Also social buffer: Target experiences TSST stressor with a friend who also experiences the stressor
- Friend Provides Support: random assignment to Friend Provides Support
  Friend Support social buffer: Target experiences TSST stressor with a friend who does NOT experience the stressor
- Unfamiliar Peer: random assignment to Unfamiliar Peer
  Unfamiliar Peer social buffer: Target experiences TSST stressor with an unfamiliar peer who also experiences the stressor
- Alone: random assignment to Alone Condition
  no social buffer: random assignment to Alone Condition
Arm/Group | Friend and Target Both | Friend Provides Support | Unfamiliar Peer | Alone
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/72 | 0/65 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/72 | 0/65 | 0/69
Other Adverse Events (participants affected / at risk) | 0/63 | 0/72 | 0/65 | 0/69

LIMITATIONS AND CAVEATS:
Note that while parents consented and completed questionnaires about their family or child, they are never the focus of analysis or considered enrolled in the study. They are consenting to their child's enrollment and reporting on their child's environment, health, and behavior.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT04311996/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04311996/ICF_001.pdf